CLINICAL TRIAL: NCT03526913
Title: Role of Platelet Rich Plasma in Enhancing Graft Take in Chronic Venous Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noha Mohsen Omar (Other)
Collaborators: Menoufia University (Other)
Responsible Party: Sponsor-Investigator, Noha Mohsen Omar, Principal Investigator, MBBCH Cairo University, Menoufia University
Organization: Menoufia University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Chronic Venous Hypertension With Ulcer and Inflammation; Chronic Ulcer of Leg or Foot
Keywords: chronic leg ulcers, PRP; split-thickness skin graft; platelet-rich plasma
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: Comparison of combined autologous PRP and skin grafting to skin grafting alone in chronic leg ulcers (comparing one ulcer to another in bilateral cases, or one half of ulcer to the other in big ulcers)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP + STSG (Experimental): autologous PRP treatments every week prior to graft placement (STSG)
  Interventions: Procedure: PRP; Procedure: STSG
- STSG Split Thickness Skin Graft (Active Comparator): skin graft (STSG) (intervention)
  Interventions: Procedure: STSG

INTERVENTIONS:
Procedure: PRP — PRP: autologous platelet-rich plasma
  Other Names: platelet rich plasma
  Arms: PRP + STSG
Procedure: STSG — skin graft: Split Thickness Skin Grafting (STSG)
  Other Names: split thickness skin graft

SUMMARY:
Chronic venous ulcers are considered a problem with a big morbidity impact on both the health facilities and patients, skin-grafting have shown not so perfect outcomes with such ulcers. In this study, the investigators compare combining autologous platelet rich plasma treatments with partial skin grafting in chronic ulcers, the results were compared to using only partial skin grafting, and among various types of chronic resistant ulcers.

DETAILED DESCRIPTION:
Fourteen patients had bilateral lower limb ulcers, and 6 of them had single large ulcers as follows; Fourteen patients with chronic venous ulcers (12 of which had bilateral ulcers, 2 had single large ulcers) Four patients, each with a single chronic post-traumatic ulcer Two patients with bilateral chronic lymphatic ulcers.

After detailed history, physical examination and investigations (such as duplex),

* Each patient with bilateral ulcers included in the study (14 patients) received treatment A on one ulcer and treatment B on the other ulcer.
* In case of patients with single large ulcers (6 patients), treatment A was done on one half of the ulcer and treatment B on the other half of the ulcer (done in ulcers with an area greater than 10 x 10 cms).
* Treatment A included pre-operative intra-lesional PRP injections in 1-week intervals for 3 times, followed by intra-operative intra-lesional injection of PRP prior to meshed graft placement. PRP was injected into the ulcer bed and ulcer edges using a sterile syringe.

Treatment B included only placement of meshed graft, with no PRP treatment.

* Pre-operative preparation: Ulcers were prepared by proper dressings and followed up until acquiring a clean bed. Debridement was done as needed to obtain clean base ready for graft placement.
* PRP preparation:

  * 10 ml of blood was drawn from each patient intra operatively (autologous PRP).
  * Blood was collected in sterile tubes, Anticoagulant Citrate Dextrose (ACD) was used for anticoagulation, which is the same substance used to preserve viable platelets in blood banks for platelet transfer.
  * Tubes were centrifuged in Beckman Allerga X-12 centrifuge for 20 mins, 3000 rpm.
  * Each 10 ml of blood yielded an average of 3-4 ml of PRP. Calcium gluconate was added in a ratio of 1:10 to PRP. Post-operative assessment was carried out by follow up clinical examination, photography and weekly biopsy samples.

ELIGIBILITY:
Inclusion criteria:

* Patients with chronic ulcers for at least 6 months.
* Age ≧ 12 years.

Exclusion criteria:

* Patients younger than 12 years of age.
* Patients with diabetes or other diseases affecting tissue healing.
* Patients with current ongoing pathologies in arterial or venous systems.
* Patients with malignant ulcers.
* Patients on corticosteroids or other drugs affecting tissue healing.
* Patients with unrealistic expectations.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Graft take | month
  percentage of graft take

CONTACTS AND LOCATIONS:
Overall Officials: Sherif M. Elkashty, PHD, Principal Investigator — Menoufia University

IPD SHARING:
Plan to Share IPD: Yes
Comparison of combined pre and intra-operative PRP treatments with STSG to only STSG in treatment of chronic ulcers with special emphasis on venous ulcers.
Supporting Information: Study Protocol
Time Frame: infinite
Access Criteria: to all researchers

REFERENCES:
- [Background] Fonder MA, Lazarus GS, Cowan DA, Aronson-Cook B, Kohli AR, Mamelak AJ. Treating the chronic wound: A practical approach to the care of nonhealing wounds and wound care dressings. J Am Acad Dermatol. 2008 Feb;58(2):185-206. doi: 10.1016/j.jaad.2007.08.048. PMID 18222318
- [Background] Raffetto JD, Khalil RA. Matrix metalloproteinases and their inhibitors in vascular remodeling and vascular disease. Biochem Pharmacol. 2008 Jan 15;75(2):346-59. doi: 10.1016/j.bcp.2007.07.004. Epub 2007 Jul 7. PMID 17678629
- [Background] Werner S, Grose R. Regulation of wound healing by growth factors and cytokines. Physiol Rev. 2003 Jul;83(3):835-70. doi: 10.1152/physrev.2003.83.3.835. PMID 12843410
- [Background] Eppley BL, Woodell JE, Higgins J. Platelet quantification and growth factor analysis from platelet-rich plasma: implications for wound healing. Plast Reconstr Surg. 2004 Nov;114(6):1502-8. doi: 10.1097/01.prs.0000138251.07040.51. PMID 15509939
- [Background] Pietramaggiori G, Scherer SS, Mathews JC, Gennaoui T, Lancerotto L, Ragno G, Valeri CR, Orgill DP. Quiescent platelets stimulate angiogenesis and diabetic wound repair. J Surg Res. 2010 May 1;160(1):169-77. doi: 10.1016/j.jss.2008.09.010. Epub 2008 Oct 10. PMID 19482315
- [Background] Kakudo N, Minakata T, Mitsui T, Kushida S, Notodihardjo FZ, Kusumoto K. Proliferation-promoting effect of platelet-rich plasma on human adipose-derived stem cells and human dermal fibroblasts. Plast Reconstr Surg. 2008 Nov;122(5):1352-1360. doi: 10.1097/PRS.0b013e3181882046. PMID 18971718
- [Background] Schultz GS, Sibbald RG, Falanga V, Ayello EA, Dowsett C, Harding K, Romanelli M, Stacey MC, Teot L, Vanscheidt W. Wound bed preparation: a systematic approach to wound management. Wound Repair Regen. 2003 Mar;11 Suppl 1:S1-28. doi: 10.1046/j.1524-475x.11.s2.1.x. PMID 12654015
- [Background] Frykberg RG, Banks J. Challenges in the Treatment of Chronic Wounds. Adv Wound Care (New Rochelle). 2015 Sep 1;4(9):560-582. doi: 10.1089/wound.2015.0635. PMID 26339534
- [Background] Knighton DR, Ciresi K, Fiegel VD, Schumerth S, Butler E, Cerra F. Stimulation of repair in chronic, nonhealing, cutaneous ulcers using platelet-derived wound healing formula. Surg Gynecol Obstet. 1990 Jan;170(1):56-60. PMID 2403699